CLINICAL TRIAL: NCT00051025
Title: A Randomized, Multicenter, Phase II Evaluation of ONTAK (Denileukin Diftitox) in Patients With Previously Treated, Indolent, B-Cell, Non-Hodgkin's Lymphoma
Brief Title: Phase II Study of ONTAK in Previously Treated Patients With Low-grade Non-Hodgkin's Lymphoma (NHL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L4389-30; NCT00005621 (obsolete NCT alias)
Record Dates: First submitted 2002-12-31; First posted 2003-01-03 (Estimated); Results first posted 2011-08-03 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Non-Hodgkin's Lymphoma; Lymphoma, B-cell; Lymphoma, Low-grade
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell | interventions — denileukin diftitox

INTERVENTIONS:
Drug: ONTAK

SUMMARY:
The purpose of this study is to look at the safety and effectiveness of ONTAK in previously treated patients with NHL.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of low-grade (indolent), B-cell, non-Hodgkin's lymphoma.
* Positive expression for CD25 of tumor cells in a lymph node biopsy as defined by greater than 20% of malignant cells staining for CD25 by standardized immunohistochemical assay.
* Modified Ann Arbor Stage I, II, III or IV.
* Patients must have received at least two but no more than five prior therapies. One prior therapy must have been cytotoxic chemotherapy and one prior therapy must have been monoclonal antibody therapy. Combination chemotherapy, including regimens used prior to bone marrow transplantation, will count as a single therapy for purposes of eligibility.
* Patients must have bidimensionally measurable disease.
* Patients must be 18 years of age or older.
* An ECOG performance status of 0, 1, or 2.
* Acceptable organ function defined as follows:

  * absolute neutrophil count (ANC) > or = to 1,000/mm3, platelet count > or = to 50,000/mm3, Hemoglobin > or = to 8 g/dL;
  * Bilirubin < or = to 1.5 times the upper limit of normal (ULN);
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < or = to 1.5 times the upper limit of normal;
  * Serum creatinine <1.8mg/dL;
  * Serum albumin > or = to 3.0 g/dL.
* New York Heart Association classification of I or II and no history of poorly controlled hypertension.
* Must be free of serious concurrent illness.
* Female patients must meet the following criteria:

  * If the patient is a female of childbearing potential, she must have negative serum beta human chorionic gonadotropin (B-hCG) pregnancy test within seven days prior to study entry and must have used an effective means of contraception or have been sexually abstinent for at least four weeks prior to the negative serum pregnancy test and through to study entry.
  * Female patients of childbearing potential must agree to practice an effective method of birth control during the entire treatment period and for at least three weeks after their last treatment on protocol.

Exclusion Criteria:

* Patients with cutaneous T-cell lymphoma.
* Patients previously treated with ONTAK (DAB389lL-2) or DAB486IL-2.
* Inability to comply with protocol requirements for this study.
* Pregnant women or lactating women who are breast feeding or women planning to become pregnant during the treatment period or three weeks after their last treatment on protocol.
* Serious intercurrent medical illnesses or active infections requiring parenteral antibiotics, which would interfere with the ability of the patient to carry out the treatment program.
* Sero-positive for human immunodeficiency virus (HIV) antibody. History of ongoing Hepatitis B or Hepatitis C infection.
* Another malignancy or history of another cancer with less than five disease-free years (other than resected basal or squamous cell skin cancers or in situ cervical cancer).
* Patients with a known hypersensitivity to ONTAK or any of its components: diphtheria toxin, interleukin-2, or excipients.
* Any investigational agents within one month prior to study entry.
* Prior radiation therapy within four weeks of enrollment or to the only site of evaluable disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2000-05; Primary Completion 2001-01 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elyane Lombardy, M.D., Study Director — Ligand Pharmaceuticals
Locations (2):
- United States (2):
  - Central Baptist Hospital, Lexington, Kentucky
  - Hematology and Oncology Services, Metairie, Louisiana

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 6 centers in U.S. during the period of 18-May-2000 to 12-May-2001
Groups:
- Ontak 4-Course Group: Four courses of Ontak 9 mcg/kg/day for 5 consecutive days every 21 days
- Ontak 8-Course Group: Eight courses of Ontak 9 mcg/kg/day for 5 consecutive days every 21 days
Period: Overall Study
Arm/Group | Ontak 4-Course Group | Ontak 8-Course Group
Started | 5 | 4
Completed | 3 | 0
Not Completed | 2 | 4
Not completed — Progressive Disease | 1 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ontak 4-Course Group | Ontak 8-Course Group | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 2 | 2 | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 65.4 (8.4) | 60.8 (15.5) | 63.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Objective Clinical Response: Complete Response (CR) or Partial Response (PR) at Week 24, or, in the Event of Lengthened Cycle Intervals, at the End of Cycle 8.
Description: Complete response: achievement of a complete regression for >4 weeks of all palpable and x-ray demonstrable disease and bone marrow disease. Partial response: response to therapy with a 75% reduction in the greatest diameters of the measurable lesions for >4 weeks and had indeterminate bone marrow biopsy
Time Frame: 24 Weeks
Population: Intent-to-treat
Measure: Number; unit: Participants
Arm/Group | Ontak 4-Course Group | Ontak 8-Course Group
Number analyzed (Participants) | 5 | 4
Participants | 1 | 1

2. Secondary Outcome: Duration of Response
Description: The duration of response was defined as the time interval from start of the first response (CR or PR) to the time of documented disease progression.
Time Frame: From beginning of response to time of relapse
Population: Intent-to-treat. Please note: Data represent 1 subject in each treatment group who responded.
Measure: Number; unit: Days
Arm/Group | Ontak 4-Course Group | Ontak 8-Course Group
Number analyzed (Participants) | 1 | 1
Days | 175 | 797

3. Secondary Outcome: Time-to-Treatment Failure
Time Frame: From start of first treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Ontak 4-Course Group | Ontak 8-Course Group
Serious Adverse Events (participants affected / at risk) | 1/5 | 1/4
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ontak 4-Course Group (N=5) | Ontak 8-Course Group (N=4)
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Chest Pain (General disorders) | 0 | 1
Progression of Mantle Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ontak 4-Course Group (N=5) | Ontak 8-Course Group (N=4)
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 2
Headache (Nervous system disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Abdominal Distention (Gastrointestinal disorders) | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 2
Lip Blister (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Asthenia (General disorders) | 1 | 1
Chest Discomfort (General disorders) | 0 | 2
Fatigue (General disorders) | 3 | 3
Oedema Peripheral (General disorders) | 2 | 1
Pain (General disorders) | 1 | 2
Pyrexia (General disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No